CLINICAL TRIAL: NCT02225535
Title: Advancing Interprofessional Primary Health Care Services in Rural Settings for People With Chronic Low Back Disorders: Investigation of a Physiotherapist and Nurse Practitioner Intervention Delivered Through Telehealth
Brief Title: Investigation of a Physiotherapist and Nurse Practitioner Intervention for Chronic Low Back Disorders Delivered Through Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); Ralston Brothers Grant (Kelsey Trail Health Region) (Unknown)
Responsible Party: Principal Investigator, Brenna Bath, Assistant Professor, School of Physical Therapy, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bio13-241
Record Dates: First submitted 2014-07-31; First posted 2014-08-26 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; telehealth; videoconferencing; access to physical therapy; interprofessional care; rural health
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (NP) (Placebo Comparator): Rural NP with client in-person, usual care
  Interventions: Other: NP face to face management of Chronic Low Back Pain
- PT in-person (Active Comparator): Urban PT travels to rural area to manage patient's back pain in-person.
  Interventions: Other: PT face to face management of Chronic Low Back Pain
- PT/NP Telehealth (Active Comparator): Intervention: Rural NP is joined by PT via Telehealth for interprofessional videoconference with patient
  Interventions: Other: Interprofessional Videoconferencing for Chronic Low Back Pain

INTERVENTIONS:
Other: NP face to face management of Chronic Low Back Pain — usual NP management of chronic low back disorder
  Arms: Usual Care (NP)
Other: PT face to face management of Chronic Low Back Pain — Includes manual therapy, education, exercise
  Arms: PT in-person
Other: Interprofessional Videoconferencing for Chronic Low Back Pain — Includes manual therapy, education, exercise.
  Arms: PT/NP Telehealth

SUMMARY:
The purpose of this project is to compare "usual care" for chronic low back disorders in a rural setting (nurse practitioner/NP) to two different means of integrating Physical Therapy (PT) into a rural health care team:

1. in-person PT assessment, where the PT travels from an urban center
2. interprofessional Telehealth assessment where the local NP is joined by a PT via Telehealth.

The project will evaluate health, systems and process outcomes, comparative effectiveness and costs of the three methods of assessment. The hypothesis is that an interprofessional Telehealth assessment with be as effective as an in-person PT assessment, but more effective than usual care.

DETAILED DESCRIPTION:
The study design will include two intervention groups and a control group with 20 participants in each group: 1. interprofessional videoconferencing intervention, 2. in-person PT and, 3. "usual-care" provided by a NP. Due to the interprofessional nature of the intervention, the NP involved in the telehealth-based intervention group may alter their "usual care" practice; therefore, the control group participants will be drawn from the practices of 2 NPs not involved in the Telehealth intervention providing services out of a different clinic. Each PT and the NP alone will complete a standardized online diagnostic classification tool.Participants will be randomly assigned to one of the three groups.

ELIGIBILITY:
Inclusion Criteria:

* adult 18-80
* low back pain and/or related leg pain affecting function, >3 months duration

Exclusion Criteria:

* clients within a third party payer insurance coverage system
* clients with primarily neck or thoracic pain
* clients with language or comprehension difficulties that would limit completion of paperwork

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Short term impact of patient/provider satisfaction | up to 2 weeks after assessment
  questionnaire
Short term outcome of patient experience with Telehealth | up to 2 weeks
  qualitative questionnaire
Medium term outcome of patient and provider satisfaction | 3 months
  questionnaire
Short term impact of patient function | up to 2 weeks after assessment
  Modified Oswestry Disability questionnaire
Short term impact on pain | up to 2 weeks after assessment
  Numeric Pain Rating Scale - questionnaire
Short term impact on quality of life | up to 2 weeks after assessment
  Euro-Qol health survey instrument (EQ-5D)
Medium term impact on pain | 3 months
  Numeric Pain Rating Scale - questionnaire
Medium term impact on quality of life | 3 months
  Euro-Qol health survey instrument (EQ-5D)
Medium impact on patient function | 3 months
  Modified Oswestry Disability Index questionnaire

SECONDARY OUTCOMES:
Cost effectiveness of each of 3 arms of study | 6 months
  patient diaries
Long term outcome on patient/provider satisfaction | 6 months
  questionnaire
Long term impact on quality of life | 6 months
  Euro-Qol health survey instrument (EQ-5D)
Long term impact on function | 6 months
  Modified Oswestry Disability Index questionnaire
Long term impact on pain | 6 months
  Numeric Pain Rating Scale

OTHER OUTCOMES:
Barriers and facilitators to use of Telehealth | 2 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Brenna Bath, PhD, Principal Investigator — School of Physical Therapy, University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Lovo S, Imeah B, Sari N, O'Connell ME, Milosavljevic S, Angarita-Fonseca A, Bath B. Effectiveness of an interprofessional assessment and management approach for people with chronic low back disorders delivered via virtual care: A randomized controlled trial pilot intervention. Digit Health. 2024 Jun 5;10:20552076241260569. doi: 10.1177/20552076241260569. eCollection 2024 Jan-Dec. PMID 38846367
- [Derived] Bath B, Lovo Grona S, Milosavljevic S, Sari N, Imeah B, O'Connell ME. Advancing Interprofessional Primary Health Care Services in Rural Settings for People with Chronic Low Back Disorders: Protocol of a Community-Based Randomized Controlled Trial. JMIR Res Protoc. 2016 Nov 9;5(4):e212. doi: 10.2196/resprot.5914. PMID 27829573